CLINICAL TRIAL: NCT05689164
Title: Long-term Follow-up Safety and Efficacy Study in Participants With Duchenne Muscular Dystrophy Who Have Received Fordadistrogene Movaparvovec in a Preceding Clinical Study
Brief Title: A Study to Understand the Long-term Safety and Effects of an Experimental Gene Therapy for Duchenne Muscular Dystrophy.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: All participants who have received fordadistrogene movaparvovec in any Pfizer study will now be assessed for long-term safety in 1 combined study: C3391003
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C3391011; NCT05689164 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Muscular Dystrophy, Duchenne; Genetic Therapy; Gene Therapy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All participants (Other): All participants enrolled in the study.
  Interventions: Biological: fordadistrogene movaparvovec

INTERVENTIONS:
Biological: fordadistrogene movaparvovec — gene therapy administered in a previous study.

SUMMARY:
The purpose of this study is to understand the safety and effects of an experimental gene therapy called fordadistrogene movaparvovec. We are seeking participants from previous Pfizer interventional studies. We will follow participants' experience in this study for 10 years after the end of their previous study. Participants will have 1 annual onsite visit and a few annual remote visits. The exact number of remote visits will be decided by their study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received fordadistrogene movaparvovec in a previous Pfizer interventional study.

Exclusion Criteria:

* Investigator site staff directly involved in the study and their family members

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with serious adverse events | At least annually from 5 through 10 years after dosing in the interventional study.
Percentage of participants with serious adverse events | At least annually from 5 through 10 years after dosing in the interventional study.
Number of participants with adverse events considered related to treatment | At least annually from 5 through 10 years after dosing in the interventional study.
Percentage of particpants with adverse events considered related to treatment | At least annually from 5 through 10 years after dosing in the interventional study
Number of participants with malignancy adverse event | At least annually from 5 through 10 years after dosing in the interventional study
Number of participants with clinically significant findings in electrocardiogram (ECG) assessments | Annually from 5 through 10 years after dosing in the interventional study.
Number of participants with clinically significant findings in cardiac troponin I laboratory examinations | Annually from 5 through 10 years after dosing in the interventional study
Number of participants with clinically significant findings in echocardiogram parameters | Annually from 5 through 10 years after dosing in the interventional study

SECONDARY OUTCOMES:
Change from pre-dose in the ability to walk 10 meters unassisted | Annually from 5 through 10 years after dosing in the interventional study.
Change from pre-dose in the ability to climb stairs. | Annually from 5 through 10 years after dosing in the interventional study
Change from pre-dose in the Performance of Upper Limb (PUL) 2.0 entry score | Annually from 5 through 10 years after dosing in the interventional study
Change from pre-dose in the North Star Ambulatory Assessment total score | Annually from 5 through 10 years after dosing in the interventional study
  Applicable to a sub-set of participants only
Change from pre-dose in percent of predicted forced vital capacity (%pFVC) and percent predicted peak expiratory flow (%pPEF) | Annually from 5 through 10 years after dosing in the interventional study
Change from pre-dose in left ventricular ejection fraction (LVEF) on echocardiogram | Annually from 5 through 10 years after dosing in the interventional study
Change from pre-dose in the Modified Pediatric Outcomes Data Collection Instrument | Annually from 5 through 10 years after dosing in the interventional study
Change from pre-dose in the Upper Limb Function Patient Reported Outcome Measure | Annually from 5 through 10 years after dosing in the interventional study
  Applicable to non-ambulatory participants only
Age when percent predicted forced vital capacity <30% | Annually from 5 through 10 years after dosing in the interventional study
Age at loss of ambulation | From 5 through 10 years after dosing in the interventional study
Age at death | From 5 through 10 years after dosing in the interventional study
Cause of death | From 5 through 10 years after dosing in the interventional study
Glucocorticoid use dose and frequency | At least annually from 5 through 10 years after dosing in the interventional study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Reed Neurological Research Center, Los Angeles, California
  - UCLA Children's Heart Center, Los Angeles, California
  - UCLA Clinical Lab Services, Los Angeles, California
  - UCLA Kameron Gait and Motion Analysis Laboratory (Westwood Rehabilitation Center), Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Duke Lenox Baker Children's, Durham, North Carolina
  - Duke Children's Health Center, Durham, North Carolina
  - University of Utah Imaging and Neurosciences Center, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - University of Utah Craig H. Neilsen Rehabilitation Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3391011